CLINICAL TRIAL: NCT01225185
Title: Assessing Cerebral Blood Flow Autoregulation in the Head-up Versus Supine Position During General Anesthesia and Its Relationship With Postoperative Neurocognitive Changes and Serum Biomarkers of Brain Injury
Brief Title: Assessing Cerebral Blood Flow Autoregulation During Surgery in the Head-up Position
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Anesthesia Patient Safety Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: APSF; 1R01HL092259 (NIH)
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Shouldersurgery
Keywords: neurological complications; brain blood flow autoregulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing shoulder surgery: This observational study will compare cerebral blood flow autoregulation in patients undergoing surgery in either the supine lateral position or the semi-recumbent or "beach chair" position. The choice of patient positioning is not randomized but based on usual surgical considerations.

SUMMARY:
Neurological injury after elective shoulder surgery in the beach chair position is thought to result from cerebral hypoperfusion and should therefore be preventable by appropriate hemodynamic monitoring and management. This proposal will use a system to continuously monitor cerebral blood flow autoregulation to identify safe arterial blood pressure targets in patients in the beach chair position, compared with a control cohort having orthopedic surgery in the lateral decubitus supine position. Autoregulation data will be compared against a new, highly specific and sensitive serum biomarker of neurologic injury, glial fibrillary acid protein, and postoperative neurocognitive testing results.

DETAILED DESCRIPTION:
Neurologic injury under general anesthesia in the beach chair position is believed to result from cerebral hypoperfusion.1 We hypothesize that brain hypoperfusion in this circumstance is caused by blood pressure monitoring that does not reflect of cerebral perfusion pressure. Maintenance of arterial blood pressure above an individual's lower limit of cerebral blood flow autoregulation would prevent this devastating complication. Near infrared spectroscopy can be used to continuously monitor autoregulation with the cerebral oximetry index (COx), a moving linear correlation coefficient between cortical tissue oxygen saturation and arterial pressure. We hypothesize that subjects in the beach chair position have impaired cerebral blood flow autoregulation compared with subjects undergoing surgery in the lateral decubitus supine position. We will test this hypothesis by comparing CBF autoregulation data, including the percentage of time patients undergoing elective surgery have abnormal autoregulation, in the beach chair position versus supine position. We will establish the range of arterial pressure required to maintain autoregulation in the two groups. Cerebral autoregulation results will be assessed for a relationship with postoperative neurocognitive dysfunction and with serum glial fibrillary acid protein levels, a biomarker of brain injury.

The specific aims of this study are:

1. To compare the average cerebral oximetry index and the percentage of time with abnormal COx between subjects in the head up or supine position during surgery under general anesthesia.
2. To compare the range of arterial blood pressure required for a normal cerebral oximetry index between subjects anesthetized in the head up or supine position.
3. To assess the association between impaired cerebral blood flow autoregulation and postoperative neurocognitive decline 1 month after surgery and perioperative elevation of serum glial fibrillary acid protein.

Monitoring autoregulation non-invasively with COx has the potential to improve patient safety by delineating individualized limits of safe ABP for patients at risk of neurologic injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older undergoing shoulder arthroscopy in the beach chair position or lateral decubitus position without elevation of the head.

Exclusion Criteria:

* Women of child bearing potential require a negative urine HCG test to be enrolled. Patients unable to attend postoperative cognitive testing sessions will be excluded from the study as will those with known allergy to adhesive tape.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 patients undergoing shoulder surgery in the supine lateral position and 120 subjects undergoing surgery in the beach chair position.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2010-07; Primary Completion 2014-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
cerebral oximetry index between subjects in the head up or supine position during surgery under general anesthesia | During surgery

SECONDARY OUTCOMES:
To compare the range of arterial blood pressure required for a normal cerebral oximetry index between subjects anesthetized in the head up or supine position. | During surgery
To assess the association between impaired cerebral blood flow autoregulation and postoperative neurocognitive decline and elevation of serum glial fibrillary acid protein. | 1 month after surgery for neurocognitive decline; perioperatively for serum GFAP levels.

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Hogue, MD, Principal Investigator — The Johns Hopkins Medical Institutions
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States